CLINICAL TRIAL: NCT06444139
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Clinical Trial to Investigate the Efficacy of Probiotics on Gastrointestinal Function in Adults With Occasional Constipation
Brief Title: Probiotic Intervention for Occasional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23PICPP01
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-11

CONDITIONS: Gut Function; Occasional Constipation
Keywords: Bowel movements; Gut function; Probiotics
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics (Active Comparator)
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics
  Arms: Probiotics
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to study the effect of probiotics on gut function in subjects with occasional constipation. The main question it aim to answer is if intake of probiotics will decrease the transit time. Participants will randomized to either consume probiotics or a placebo product.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 - 65 years
* With occasional constipation
* Agrees to maintain current lifestyle habits
* Healthy
* Provided voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
* Allergy, sensitivity, or intolerance to study products or clinical assessment materials
* Chronic constipation
* Current or history of significant diseases or abnormalities of the gastrointestinal tract (examples (include but are not limited to atrophic gastritis, celiac disease, gluten intolerance/sensitivity, inflammatory bowel disease)
* Unstable metabolic disease or chronic diseases
* Unstable hypertension.
* Type I or Type II diabetes, cancer
* Significant cardiovascular event in the past 6 months. History of or current diagnosis with kidney and/or liver diseases
* Self-reported confirmation of current or pre-existing thyroid condition.
* Individuals with an autoimmune disease or are immune compromised
* Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis, blood/bleeding disorders
* Any other condition or lifestyle factor, that may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Transit time | Baseline to day 56
  Difference in change in gut transit time as assessed by blue-dye method

SECONDARY OUTCOMES:
Bowel movements | Baseline to day 28 and day 56
  Frequency of complete and spontaneous bowel movements (CSBM)
Stool consistency | Baseline to day 28 and day 56
  Evaluated by Bristol stool form scale
Bloating and flatulence | Baseline to day 28 and day 56
  Frequency
Quality of life | Baseline to day 28 and day 56
  Evaluated by a questionnaire
Digestive symptoms | Baseline to day 28 and 56
  Evaluated by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Science Clinic, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No